CLINICAL TRIAL: NCT06703047
Title: Tislelizumab Combined with Chemotherapy and All Trans Retinoic Acid for Locally Advanced or Metastatic Esophageal Squamous Cell Carcinoma: a Prospective, Double-blind, Multicenter, Randomized Controlled Phase II Trial
Brief Title: Tislelizumab Combined with Chemotherapy and All Trans Retinoic Acid for Locally Advanced or Metastatic Esophageal Squamous Cell Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Yu hui, Chief physician, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ESCC-ATRA-IIT-01
Record Dates: First submitted 2024-10-23; First posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- All trans tretinoic acid+tislelizumab+chemotherapy (paclitaxel, cisplatin, or carboplatin) (Experimental)
  Interventions: Drug: ATRA+pd-1+chemo
- Placebo+tislelizumab+chemotherapy (paclitaxel, cisplatin, or carboplatin) (Placebo Comparator)
  Interventions: Drug: placebo+PD-1+chemo

INTERVENTIONS:
Drug: ATRA+pd-1+chemo — All trans tretinoic acid+tislelizumab+chemotherapy (paclitaxel, cisplatin, or carboplatin)
  Arms: All trans tretinoic acid+tislelizumab+chemotherapy (paclitaxel, cisplatin, or carboplatin)
Drug: placebo+PD-1+chemo — Placebo+tislelizumab+chemotherapy (paclitaxel, cisplatin, or carboplatin)
  Arms: Placebo+tislelizumab+chemotherapy (paclitaxel, cisplatin, or carboplatin)

SUMMARY:
Tislelizumab combined with chemotherapy and all trans retinoic acid for locally advanced or metastatic esophageal squamous cell carcinoma: a prospective, double-blind, multicenter, randomized controlled phase II trial

DETAILED DESCRIPTION:
This study is a prospective, double-blind, multicenter, randomized controlled phase II clinical trial of tislelizumab combined with chemotherapy and all trans retinoic acid in the treatment of locally advanced non-surgical or metastatic esophageal squamous cell carcinoma. The aim is to evaluate the efficacy and safety of tislelizumab combined with chemotherapy and all trans retinoic acid in the treatment of locally advanced non-surgical or metastatic esophageal squamous cell carcinoma. Patients with locally advanced inoperable or metastatic ESCC can only be enrolled after meeting the criteria. They will receive treatment with tislelizumab combined with chemotherapy+all trans retinoic acid or tislelizumab combined with chemotherapy+placebo, with a treatment cycle of every 3 weeks. The treatment will continue until disease progression or reaching the criteria for terminating the study drug treatment, for a maximum of two years.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects voluntarily participate and sign a written informed consent form;
2. Age ≥ 18 years old;
3. Diagnosed by pathological histology as an inoperable locally advanced or metastatic esophageal squamous cell carcinoma patient;
4. According to AJCC 8th edition staging and RECIST 1.1 solid tumor evaluation criteria, there must be at least one measurable lesion;
5. Have not received any local or systemic anti-tumor treatment for locally advanced/metastatic esophageal squamous cell carcinoma. For patients who have received adjuvant/neoadjuvant chemotherapy, or radical radiotherapy for advanced diseases, if there is a gap of at least 6 months between disease progression or recurrence and the end of the last drug treatment, they are allowed to be included in this study;
6. The main organs function is good;
7. Expected survival period ≥ 3 months;
8. ECOG PS score: 0-1 points;
9. According to the researcher's judgment, the patient has the ability to follow the research protocol.
10. Non surgical sterilization or female patients of childbearing age are required to use a medically approved contraceptive measure (such as intrauterine device, contraceptive pill, or condom) during the study treatment period and within 6 months after the end of the study treatment period; Female patients of childbearing age who undergo non-surgical sterilization must have a negative serum or urine HCG test within 72 hours prior to enrollment in the study; And it must be during non lactation period; For male patients whose partners are women of childbearing age, effective contraception methods should be used during the trial period and within 6 months after the last dose.

Exclusion Criteria:

1. Patients who have received immunotherapy;
2. Individuals who are allergic to the drugs or their components used in this study;
3. The patient currently (within 3 months) has digestive tract diseases such as esophageal varices, active ulcers of the stomach and duodenum, ulcerative colitis, portal hypertension, or other conditions determined by the researchers that may cause gastrointestinal bleeding or perforation;
4. There are small cell carcinoma, adenocarcinoma, or mixed cancer components in histology;
5. Central nervous system metastasis has occurred;
6. Complete esophageal obstruction;
7. Unable to tolerate gastrointestinal endoscopic biopsy; Having clear concerns about gastrointestinal bleeding (such as local active ulcer lesions, positive fecal occult blood); History of gastrointestinal bleeding within 6 months;
8. Patients with primary malignant tumors other than esophageal cancer (excluding cured skin basal cell carcinoma and cervical carcinoma in situ);
9. Existence of any active autoimmune disease or history of autoimmune disease with expected recurrence;
10. Discovering a high risk of esophageal fistula through clinical evaluation or imaging examinations, such as a history or related symptoms of esophageal fistula, or primary tumor infiltration into large blood vessels or trachea;
11. If patients with uncontrolled tumor related pain require analgesic treatment, the treatment plan used at the time of enrollment in the study must be stable;
12. Individuals who tested positive for HIV during screening;
13. Individuals who test positive for hepatitis C virus (HCV) during screening;
14. HBV positive and cccDNA ≥ 500 IU/mL during screening;
15. Within the 6 months prior to enrollment, have any of the following diseases: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass surgery, symptomatic congestive heart failure, or cerebrovascular accident;
16. Pregnant or lactating women or those who have the ability to conceive but have not taken contraceptive measures;
17. Individuals with other serious acute or chronic physiological or mental problems;
18. Participated in any other drug clinical studies within 4 weeks prior to the first administration

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-11-20 (Estimated); Primary Completion 2029-11-20 (Estimated); Study Completion 2030-10-24 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | up to 3 years

SECONDARY OUTCOMES:
Objective Response Rate | up to 3 years
Progression Free Survival | up to 3 years
Disease control rate | up to 3 years
Duration of Response | up to 3 years
Single cell TCR sequencing, whole exome sequencing, RNA seq, and methylation sequencing were performed on tumor tissue and blood samples | up to 3 years
Skin adverse reactions | up to 3 years
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | up to 3 years
EORTC QLQ-30 | up to 3 years
EORTC QLQ-LC13 | up to 3 years

IPD SHARING:
Plan to Share IPD: No